CLINICAL TRIAL: NCT03372252
Title: Impact of the Inspiratory Cortical Control on the Outcome of the Ventilatory Weaning Test in Patients Intubated in Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BRAIN-WEAN
Record Dates: First submitted 2017-09-23; First posted 2017-12-13 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Respiration Disorder; Respiratory Failure; Weaning Failure; Respiratory Compensation; Respiratory Center Dysfunction
MeSH Terms: conditions — Respiration Disorders; Respiratory Insufficiency | interventions — Electroencephalography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Successful weaning (Experimental): Patients extubated after the success of the breathing test in spontaneous ventilation under artificial nose and always extubated after seven days.
  Interventions: Device: Electroencephalography
- Failure to wean (Experimental): Patients who failed the breathing test in spontaneous ventilation under artificial nose and not extubated or patients extubated after the success of the weaning test in spontaneous ventilation under artificial nose but reintubated within seven days.
  Interventions: Device: Electroencephalography

INTERVENTIONS:
Device: Electroencephalography — Simplified electroencephalography using three electroencephalogram electrodes and two electro-oculogram electrodes for the measurement of central respiratory control through the inspiratory premotor potentials.

SUMMARY:
In case of respiratory distress, patients are intubated to be connected to an artificial respirator to ensure gas exchanges. Before any ventilatory weaning, a breathing test in spontaneous ventilation under artificial nose is practiced. The patient keeps the endotracheal tube but is no longer assisted by the ventilator. Mortality is markedly increased with the prolongation of the weaning period. Despite the presence of all weaning criteria and the success of a breathing test in spontaneous ventilation under artificial nose, failure of extubation occurs in 20% of patients.

Experimental application of an additional inspiratory load in awake healthy subjects causes a compensatory increase in respiratory work to maintain effective ventilation, and the subject does not develop hypoventilation. This respiratory drive to breathe has been demonstrated by quantified electroencephalography in inspiratory load tests in the form of pre-inspiratory negative deflections of low amplitude similar to the potential described during the preparation of the voluntary movement of a limb. These inspiratory pre-motor potentials begin about 2.5 seconds before the start of a movement in the additional motor area.

Does the simple and noninvasive analysis of inspiratory cortical control during the spontaneous ventilation breath test under artificial nose predict the outcome of this test as well as weaning at 7 days?

ELIGIBILITY:
Inclusion Criteria:

* All intubated-ventilated patients eligible for an artificial nose breathing test in spontaneous ventilation, according to the physician in charge, and to the protocol of the medical resuscitation service and good clinical practice,
* at least 18 years of age;
* intubated-ventilated for at least 24 hours;
* express consent given by patients or "relatives" after clear and fair information on the study.

Exclusion Criteria:

* Patients are secondarily excluded from the study only if EEG or pressure monitoring are uninterpretable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- university hospital center of Poitiers, Poitiers, Vienne, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 patients included but 62 patients could have been analyzed for technical maters
Groups:
- SBT Success: 45 patients (73%) succeded the Spontaneous breathing trial
- SBT Failure: 17 patients (27%) failed the Spontaneous breathing trial
Period: Overall Study
Arm/Group | SBT Success | SBT Failure
Started | 45 | 17
Completed | 45 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SBT Success | SBT Failure | Total
Number analyzed (Participants) | 45 | 17 | 62
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [56 to 67] | 70 [62 to 76] | 63 [57 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 5 | 25
  Male | 25 | 12 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Median (Inter-Quartile Range); unit: kg/m²] | 30 [26 to 34] | 32 [28 to 34] | 31 [27 to 34]

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of Inspiratory Premotor Potentials
Description: Amplitude in microvolts of the inspiratory premotor potentials measured during the first 15 minutes of the artificial noses breathing test in patients who successfully passed their ventilatory withdrawal and in patients who failed their withdrawal.
Time Frame: Fifteen minutes
Measure: Median (Inter-Quartile Range); unit: µV
Arm/Group | SBT Success | SBT Failure
Number analyzed (Participants) | 45 | 17
µV | 1.2 [0.5 to 2.0] | 2.1 [1.7 to 2.9]

ADVERSE EVENTS:
Time Frame: from enrollement until the end of the spontaneous breathing trial the same day for the primary objective's mesurement and until 7 days for the whole follow up.
Arm/Group | SBT Success | SBT Failure
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/17
Other Adverse Events (participants affected / at risk) | 0/45 | 0/17

LIMITATIONS AND CAVEATS:
Patients were not consecutively recruited due to the limited availability of investigator/research materials followed by the COVID- 19 pandemic. As a result, this study presents only a fraction of the eligible population. PIP methodology is complex and requires EEG recording and sophisticated EEG signal analysis, which was performed off-line in our study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT03372252/Prot_SAP_000.pdf